CLINICAL TRIAL: NCT05329467
Title: Validation of Pain Assessment Tool FTS
Brief Title: Validation of Pain Assessment Scale Faces Thermometer Scale (FTS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lund University (Other)
Collaborators: Jonkoping University (Other); Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PR2020-0026
Record Dates: First submitted 2021-11-10; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Pain; Assessment, Self; Child, Only
Keywords: validation
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Validation (Other)
  Interventions: Other: Validation of Faces Thermomether Scale

INTERVENTIONS:
Other: Validation of Faces Thermomether Scale — Participants are introduced to all three painscales and are asked to rate their pain with each and one of them according to instructions for each scale

SUMMARY:
The aim of the study was to psychometrically evaluate the electronic self assessment Faces Pain Scale (FPS). Validation is performed in relation to golden standard of pain scale assessments Faces Pain Scale Reversed (FPS-R) and Coloured analogue Scale (CAS). 600 children with a range of illnesses on various paediatric healthcare settings in Sweden, Island, Denmark and USA will be included. Pain assessment will take place postoperatively, in relation to procedures or in a setting where acute pain is identified.

DETAILED DESCRIPTION:
The Faces Pain Scale-Revised (FPS-R) and Coloured Analogue Scale (CAS), two commonly used analogue pain scales for self-report with good validity and reliability in psychometric evaluations with children 8-17 years of age were used as golden standard for study 1. A systematic review found strong recommendation for the use of FPS-R and CAS for acute pain and weak endorsement for post-operative pain in children above the age of seven9.

Procedure A convenience sample of total of 600 children 8-17 years of age will be enrolled in four groups with 150 children in each group based on a power calculation Group 1: Children with no pain. Group 2: Children experiencing acute pain requiring pain treatment/pain management. Group 3: Children who will undergo medical procedures that are associated with pain, e.g., intramuscular injections, lumbar punctures, and wound care awakening and without strong sedatives. Group 4: Children who will undergo minor surgery. The data collection follows a predetermined study protocol, estimated time for data collection is six to twelve months at each site to fulfil power calculation requisites. Prior to data collection, a pilot study will be done with children (n=20) at Skåne University Hospital and the study protocol will be evaluated for cultural sensitivity with children (n=5) in each country. All assessments will be performed in the child's primary language. In all encounters the words "hurt" or "pain" will be used interchangeably, depending on what seem to be most understandable for each child. The attending nurse/physician will identify eligible study participants and provides the child and the child's caregivers with oral and written information about the study and seeks formal informed consent. The child will be allocated a personal study code. The code also determines the randomized order of pain assessment, i.e., FTS→FPS-R→CAS; CAS→FTS→FPS-R; FPS-R→CAS→FTS which will be used for all assessments by the child to avoid assessment bias. The nurse will present each of the three scales to the child in the same order as assigned to the particular child for the assessment. Data on pain assessment will be collected at specific time points according to which of the four groups it is (Figure 4).

Data from the digital FTS assessment will be transformed by the nurse and documented together with data from FPS-R and CAS into a coded individual paper study form. At all follow- up assessments the child will be asked if he/she experiences more, less, or about the same level of pain as at the previous assessment.

Psychometric properties in terms of validity and reliability of the FTS in relation to the FPS-R and the CAS in our study population will be determined by the use of comparative statistics. Most adequate tests (e.g., Pearson's or Spearman's correlation, regression analysis) will be chosen s depending on data distribution. For group 1 a cut-off score at 0-3 and for group 2 cut-off at 4-10 will be used.

Convergent validity will be assessed by determining correlations and agreement between the FTS, the FPS-R and the CAS for self-assessing pain in children. Discriminative validity (being part of convergent validity) will be assessed to determine to what extent the FTS actually measure only the construct pain, and not something else (e.g., anxiety) by comparing the initial mean FTS, FPS-R, and CAS scores in children with painful conditions, versus those with non-painful conditions. Construct validity (responsivity) in children with painful conditions will be determined by comparing the initial mean FTS, FPS-R, and CAS pain scores with their respective post-treatment pain score. Children with no pain will be assessed in a similar fashion and expect that there should be no difference between the initial and 30-45-minute scores. Reliability (the degree to which pain scores are consistent from one assessment to the next) will be assessed by test-retest analysis in the subgroup of children with painful conditions reporting that their pain is "about the same" both pre- and post-treatment.

Demographic data, e.g., age, sex, native spoken language and ethnicity will be collected through a questionnaire filled out by the child or caregiver. Data on diagnosis, reason for care and information on pain management between assessment one and two, will be collected through a questionnaire in the study form filled out by the nurse. Study forms will be collected from the site by the research group (local PI at each site) and transformed and stored at a secure digital database at Lund University.

Pain assessment will be performed two - four times each with all three scales. Their ratings are documented digitally via the FTS Webb browser on the tablet that provides the scale and by the analogous on a study protocol by the nurse for the two analogue scales. The children provide background data on a questionnaire at baseline. Consecutive sampling will be performed to include another 100 children in 8-17 for evaluation of anticipated pain by the use of the Charleston Paediatric Pain Pictures (CPPP). The child is asked to grade the anticipated level of pain that they associate the illustration on each picture with. The researcher will encourage the child to describe how they reach their decision using a "think-aloud" method. The child's reasoning will be recorded and transcribed verbatim and analysed using a phenomenographic method.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8-17
* Typically developed child
* Child and caregiver with the ability to understand spoken Swedish

Exclusion Criteria:

• Children with unstable disease or in need of ICU

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2021-09-17 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Faces Thermometer Scale validity | Change in pain assessment at up to 4 hours
  The Faces Thermometer Scale is a digital pain measure tool, which allows individuals to rate pain experience on a scale from 0 to 10. A higher reading indicates higher pain intensity.

SECONDARY OUTCOMES:
Faces Thermometer Scale content validity validity | Change in pain assessment at up to 4 hours
  The Faces Thermometer Scale is a digital pain measure tool, which allows individuals to rate pain experience on a scale from 0 to 10. A higher reading indicates higher pain intensity.
Color Analog Scale validity | Change in pain assessment at 4 hours
  The Color Analog Scale is an analog pain measure tool, which allows individuals to rate pain experience on a scale on a continuous scale which for the observer corresponds to a scale from 0 to 10 at intervals of 0.25. A higher reading indicates higher pain intensity.
Faces Pain Scale-Revised validity | Up to 15 min
  The Faces Pain Scale-Revised is an analog pain measure tool, which allows individuals to rate pain experience on a scale from 0 to 10 at intervals of 2. A higher reading indicates higher pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: charlotte castor, phd, Principal Investigator — Lund University
Locations (2):
- Sweden (2):
  - Universitetssjukhuset i Linköping, Linköping
  - Skåne University Hospital, Lund

IPD SHARING:
Plan to Share IPD: Yes